CLINICAL TRIAL: NCT05985213
Title: Cohort Study of Inpatients and Outpatient Patients With Cerebral Small Vessel Disease
Status: Recruiting | Type: Observational
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-128
Record Dates: First submitted 2023-05-25; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Small Vessel Diseases
MeSH Terms: conditions — Cerebral Small Vessel Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Each patient will provide 2 tubes of fasting blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CSVD patients: The neuroimaging diagnosis will follow the Standards for Reporting Vascular Changes on Neuroimaging (STRIVE) criteria established by the neuroimaging experts in 2013. The interpretation and assessment will be conducted jointly by one experienced radiologist and one experienced neurologist.
  Interventions: Other: data collection and follow-up

INTERVENTIONS:
Other: data collection and follow-up — Main measures and data collection methods:
  1. Recording of baseline demographic and clinical information of the participants.
  2. Multimodal magnetic resonance imaging
  3. blood pressure variability.
  4. neuropsychological testing
  5. Blood samples collection

SUMMARY:
This cohort study involves the dynamic collection of clinical information, including serum parameters , blood pressure variability, imaging data, and neuropsychological scales, in patients with cerebral small vessel disease (CSVD). The study aims to summarise the clinical and imaging characteristics of the CSVD population and identify novel CSVD risk factors. Additionally, this study intend to uncover the mechanisms underlying the clinical and imaging outcomes of CSVD. Furthermore, a multivariable prediction model for cognitive and mood disorders in patients with CSVD will be established.

DETAILED DESCRIPTION:
Research Objectives:

1. To conduct a longitudinal study on patients with cerebral small vessel disease (CSVD) and observe the dynamic evolution of their cognitive functioning, emotional disorders, and other related factors.
2. To explore and summarize the clinical and radiological characteristics of the CSVD population, and identify new risk factors for CSVD.
3. To investigate in depth the underlying mechanisms and the relationship between clinical and radiological outcomes in CSVD.
4. To establish a multifactor prediction model for cognitive and emotional disorders in CSVD.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged between 18 and 80 years, with no restriction on gender.
2. Participants who have completed a 3.0T MRI of the head within one year at Yueyang Hospital, and meet the imaging diagnostic criteria of the 2013 STRIVE guidelines.
3. Participants who have a Modified Rankin Scale (mRS) score of 0-2 (able to perform activities of daily living) at the time of the visit.
4. Participants who are able to understand and agree to participate in the study, and have signed the informed consent form.

Exclusion Criteria:

1. Diagnosis of symptomatic lacunar syndrome without 6 months of onset (participants can be enrolled after 6 months to avoid the impact of the acute phase).
2. Intracranial and extracranial vascular examination confirms stenosis of the blood vessel by ≥50%.
3. Imaging data reveals intracranial space-occupying lesions.
4. A history of other neurological or mental illnesses with a definite diagnosis of the cause, including stroke (excluding lacunar infarctions), neurodegenerative diseases (such as Parkinson's disease and Alzheimer's disease).
5. Co-occurring serious illnesses, such as malignant tumors, heart failure, respiratory failure, renal failure, severe liver dysfunction, severe blood system diseases, or gastrointestinal bleeding.
6. Severe impairment in vision, hearing, language function, or limb muscular weakness that prevents completion of relevant tests.
7. Women who are pregnant or breastfeeding.
8. MRI scan contraindicated due to various reasons (such as claustrophobia).
9. Any other reasons that prevent the collection of clinical data required for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with CSVD
Sampling Method: Non-Probability Sample
Enrollment: 1078 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive state | 2020-12-1 to 2027-12-31
  The cognitive function assessment based on Montreal Cognitive Assessment(MoCA) scale.

SECONDARY OUTCOMES:
Blood pressure variability | 2020-12-1 to 2027-12-31
  24-hour ambulatory blood pressure
The development of white matter hyperintensities, microbleeds, lacunes and, perivascular spaces. | 2020-12-1 to 2027-12-31
  If the fine structures are not clearly visible on the 3.0T MRI and further evaluation is needed for the clinical and therapeutic assessment of cerebral small vessel disease, the patient will be referred to undergo a 7.0T MRI examination.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No